CLINICAL TRIAL: NCT00150046
Title: A 12-month, Multicenter, Randomized, Open-label Non-inferiority Study of Renal Function and Efficacy Comparing Concentration-controlled Certican (1.5 mg/Day Starting Dose) With Reduced Neoral Dose Versus MMF With Standard Neoral Dose in de Novo Heart Transplant Recipients
Brief Title: Efficacy and Safety of Everolimus in de Novo Heart Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRAD001A2411
Record Dates: First submitted 2005-08-26; First posted 2005-09-08 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2011-11

CONDITIONS: Heart Transplantation
Keywords: Heart transplantation; Everolimus; Heart transplant recipient
MeSH Terms: interventions — Everolimus

INTERVENTIONS:
Drug: Everolimus

SUMMARY:
This study will test the safety and efficacy of everolimus on heart transplant recipients.

This study is not recruiting in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Male or female cardiac recipients 18-65 years of age undergoing primary heart transplantation. The graft must be functional at the time of randomization.
* Calculated creatinine clearance (Cockroft-Gault) ≥ 50 mL/min at screening.
* Patients who have given written informed consent to participate in the study.

Exclusion Criteria:

Patients who are recipients of multiple solid organ transplants or have previously received organ transplants.

Patients who received any investigational drug or who have been treated with an immunosuppressive drug or treatment within 1 month prior to randomization Patients receiving induction therapy which is not standard per local practice Patients with donor greater than 60 years and/or with known donor coronary or heart disease at the time of transplant.

Donor heart cold ischemic time >6 hours. Patients with Panel Reactive Antibodies >20%. Patients who are recipients of ABO incompatible transplants Patients with platelet count <50,000/mm3 at the evaluation before randomization.

Presence of severe hypercholesterolemia (≥350 mg/dL; ≥9 mmol/L) or hypertriglyceridemia (≥750 mg/dL; ≥8.5 mmol/L) Patients with an absolute neutrophil count of ≤1,500/mm3 or white blood cell count of ≤4000/mm3 at baseline before surgery Patients with a history of significant coagulopathy or medical condition requiring long term anti-coagulation after transplantation (low dose aspirin treatment is allowed) Patients who are HIV-positive or Hepatitis C (PCR+ only) or B surface antigen positive. Laboratory results obtained within 6 months prior to study entry are acceptable.

Recipients of organs from donors who test positive for Hepatitis B surface antigen or Hepatitis C (PCR+ only) are excluded Patients with a known hypersensitivity to similar drugs and to the components of the formulations Patients being treated with terfenadine, astemizole, or cisapride. Patients who are treated with drugs strong inducers or inhibitors of cytochrome P450 3A4.

Patients with any past (within the past 5 years) or present malignancy (other than excised basal cell carcinoma) Patients with clinically significant systemic infection Patients who are unable to take oral medication Existence of any surgical or medical condition, which in the opinion of the investigator, might significantly alter the absorption, distribution, metabolism and excretion of study medication, and/or the presence of severe diarrhea or active peptic ulcer Abnormal physical or laboratory findings of clinical significance within 2 weeks of randomization which would interfere with the objectives of the study Females of childbearing potential who are planning to become pregnant, who are pregnant and/or lactating, who are unwilling to use effective means of contraception

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2004-12; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
compare renal function

SECONDARY OUTCOMES:
compare rates of acute rejection, efficacy and safety

CONTACTS AND LOCATIONS:
Overall Officials: Basel Novartis Pharma AG, Study Chair — Basel Novartis Pharma AG
Locations (2):
- Novartis Investigational Site, Germany, Germany
- Basel Novartis Pharma AG, Basel, Switzerland

REFERENCES:
- [Result] Lehmkuhl et al., Transplantation, Volume 88, Number 1, July 15, 2009
- [Derived] Vigano M, Dengler T, Mattei MF, Poncelet A, Vanhaecke J, Vermes E, Kleinloog R, Li Y, Gezahegen Y, Delgado JF; RAD A2411 Study Investigators. Lower incidence of cytomegalovirus infection with everolimus versus mycophenolate mofetil in de novo cardiac transplant recipients: a randomized, multicenter study. Transpl Infect Dis. 2010 Feb;12(1):23-30. doi: 10.1111/j.1399-3062.2009.00448.x. Epub 2009 Sep 9. PMID 19744284